CLINICAL TRIAL: NCT00191659
Title: A Randomised, Controlled, Open-Label Study of the Broader Efficacy of Atomoxetine Hydrochloride in the Treatment of Attention-Deficit/Hyperactivity Disorder (ADHD) in Children and Adolescents
Brief Title: Study of Broader Efficacy of Atomoxetine in the Treatment of ADHD in Children/Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6962; B4Z-BP-LYBS
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-03-02 (Estimated); Status verified 2007-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Atomoxetine Hydrochloride

SUMMARY:
To test the hypothesis that children/adolescents with ADHD, who are treated with atomoxetine hydrochloride in comparison to standard current therapies have greater improvements in their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD

Exclusion Criteria:

* Patients who weigh less than 20kg at visit 1
* Have Bipolar Disorder/seizure disorder/taken anticonvulsants for seizures
* Judged to be at suicidal risk
* Taking psychotropic medication on a regular basis
* Hypertension

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200
Dates: Start 2004-06; Study Completion 2006-04

PRIMARY OUTCOMES:
To test whether atomoxetine given for 10 weeks is superior to standard current therapy as measured by CHIP-CE (Child Health and Illness Profile - Child Edition)

SECONDARY OUTCOMES:
CHIP-CE total mean score after 4 weeks of treatment.
The domains of the CHIP-CE after 4 and 10 weeks of treatment.
The following are measured after both 4 and 10 weeks of treatment:
Family Buden of Illness
Harter Self Perception Profile
ADHD-RS
Clinical Global Impression- Severity
Clinical Global Impression -Improvement
To assess whether changes to the above scales are maintained over long term
Long-term safety of atomoxetine

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559), Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Basingstoke, Hampshire, United Kingdom

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com